CLINICAL TRIAL: NCT02885805
Title: Sun Protection Factor (SPF) Efficacy Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18322
Record Dates: First submitted 2016-08-03; First posted 2016-09-01 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF evaluation + Control (Experimental): Fair-skinned subjects in good health with Skin Types I, II or III.
  Interventions: Drug: BAY987516; Drug: SPF 15 Control

INTERVENTIONS:
Drug: BAY987516 — 2.00 mg/cm2 ± 0.04 mg/cm2
Drug: SPF 15 Control — 2.00 mg/cm2 ± 0.04 mg/cm2

SUMMARY:
Evaluation of the effectiveness of a sunscreen product by determining its Sun Protection Factor (SPF) on the skin of human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I, II and/or 111 for UVB testing; Fitzpatrick Skin Type II, 111 and/or IV for UVA testing.
* Sex: Male or female.
* Age: 18-70 years.
* Good health as determined from the HRL SHF.
* Signed and dated lnformed Consent Form.
* Signed and dated HIPAA Form.
* An unambiguous MED or MPPD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Sun Protection Factor (SPF) efficacy on the skin of human subjects before a total of 2 hours of water Immersion | up to 24 hours post-exposure
  The subsites on each of the protected test sites [test sunscreen and/or Control] shall be exposed to UV light. The value of each subsite exposure shall be as appropriate to the test Method: the subject's Minimal Erythema Dose (MED) or MPPD Minimal Persistent Pigment Darkening Dose (MPPD) multiplied by the specific time intervals required. The unprotected skin site is divided into five subsites and shall also be exposed to UV light. The time intervals selected are a geometric series represented by (1.25)n, (n = the subjects MED or MPPD, at the middle [3"'] subsite) wherein each exposure time interval is 25 percent greater than the previous time or intensity. The SPF of each TM for each subject is then calculated from the exposure time interval required to produce the MED or MPPD of the protected skin, and from the exposure time interval required to produce the MED or MPPD of the unprotected skin.
Sun Protection Factor (SPF) efficacy on the skin of human subjects after a total of 2 hours of water Immersion | up to 24 hours post-exposure
  The subsites on each of the protected test sites [test sunscreen and/or Control] shall be exposed to UV light. The value of each subsite exposure shall be as appropriate to the test Method: the subject's Minimal Erythema Dose (MED) or MPPD Minimal Persistent Pigment Darkening Dose (MPPD) multiplied by the specific time intervals required. The unprotected skin site is divided into five subsites and shall also be exposed to UV light. The time intervals selected are a geometric series represented by (1.25)n, (n = the subjects MED or MPPD, at the middle [3"'] subsite) wherein each exposure time interval is 25 percent greater than the previous time or intensity. The SPF of each TM for each subject is then calculated from the exposure time interval required to produce the MED or MPPD of the protected skin, and from the exposure time interval required to produce the MED or MPPD of the unprotected skin.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Union, New Jersey, United States